CLINICAL TRIAL: NCT00654290
Title: Effect of Prophylaxy of Amiodarone and Propranolol and Amiodarone With Propranolol in Prevention of Atrial Fibrillation Post Coronary Artery Bypass Graft, A Prospective Double-Blind Randomized Study
Brief Title: Effect of Prophylaxy of Amiodarone and Propranolol and Amiodarone With Propranolol in Prevention of Atrial Fibrillation Post Coronary Artery Bypass Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: shiraz university of medical sciences/Dr kojuri, National Institute of Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 55318; NIH of IRAN
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; coronary bypass; Amiodarone; Propranolol; Coronary Artery Bypass Graft (CABG)
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone; Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- P (Experimental): Propranolol from 7 days pre-operation to 5 days post CABG
  Interventions: Drug: Propranolol
- A (Active Comparator): Amiodarone treated 7 days pre-operation to 5 days post CABG
  Interventions: Drug: Amiodarone
- AP (Active Comparator): Amiodarone and Propranolol 7 days pre-operation to 5 days post CABG
  Interventions: Drug: Amiodarone + Propranolol

INTERVENTIONS:
Drug: Amiodarone + Propranolol — Amiodarone and Propranolol 7 days pre-operation to 5 days post CABG
  Arms: AP
Drug: Amiodarone — Amiodarone treated 7 days pre-operation to 5 days post CABG
  Arms: A
Drug: Propranolol — Propranolol from 7 days pre-operation to 5 days post CABG
  Arms: P

SUMMARY:
Atrial fibrillation is the most common arrhythmia post coronary bypass surgery, currently B-blockers are the class I indication to prevent AF post CABG. We decide to evaluate use of propranolol and amiodarone separately and together to find a better prophylaxis for AF peri-CABG

DETAILED DESCRIPTION:
In this double blind randomized study 240 consecutive patients underwent elective coronary artery bypass grafting, being randomized prospectively into three groups, propranolol (p) (n=80), amiodarone (A) (n=80) and amiodarone with propranolol (AP) (n=80).

All groups received their medications from 7 days preoperatively and continued their medications for 5 days post CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patient who are going to have elective CABG
* Signing informed consent

Exclusion Criteria:

* EF<35%
* Bradycardia<60 per min
* Hypotension< 100 mmhg

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
incidence of atrial fibrillation post CABG | 7 days post CABG

SECONDARY OUTCOMES:
bradycardia, mortality, hypotension, morbidity | 7 days post CABG

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences/Cardiac Surgery and Cardiology Ward/Namazi and Shahid Faghihi Hospital, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Kojuri J, Mahmoodi Y, Jannati M, Shafa M, Ghazinoor M, Sharifkazemi MB. Ability of amiodarone and propranolol alone or in combination to prevent post-coronary bypass atrial fibrillation. Cardiovasc Ther. 2009 Winter;27(4):253-8. doi: 10.1111/j.1755-5922.2009.00100.x. PMID 19903189